CLINICAL TRIAL: NCT01822509
Title: A Phase I/IB Study of Ipilimumab or Nivolumab in Patients With Relapsed Hematologic Malignancies After Allogeneic Hematopoietic Cell Transplantation
Brief Title: Ipilimumab or Nivolumab in Treating Patients With Relapsed Hematologic Malignancies After Donor Stem Cell Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00739; NCI-2013-00739 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 12-537; 9204 (Other: Dana-Farber Cancer Institute); 9204 (Other: CTEP); P30CA006516 (NIH); R01CA183559 (NIH); U01CA062490 (NIH); UM1CA186709 (NIH)
Record Dates: First submitted 2013-04-01; First posted 2013-04-02 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplant Recipient; Myeloproliferative Neoplasm; Recurrent Acute Lymphoblastic Leukemia; Recurrent Acute Myeloid Leukemia; Recurrent Chronic Lymphocytic Leukemia; Recurrent Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Recurrent Hematologic Malignancy; Recurrent Hodgkin Lymphoma; Recurrent Myelodysplastic Syndrome; Recurrent Non-Hodgkin Lymphoma; Recurrent Plasma Cell Myeloma
MeSH Terms: conditions — Myeloproliferative Disorders; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Hematologic Neoplasms; Hodgkin Disease; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Multiple Myeloma | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ipilimumab, nivolumab) (Experimental): See Detailed Description.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Biological: Nivolumab

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; Ipilimumab Biosimilar CS1002; MDX-010; MDX-CTLA4; Yervoy
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo

SUMMARY:
This phase I/Ib trial studies the side effects and best dose of ipilimumab or nivolumab in treating patients with cancers of the blood and blood-forming tissues (hematologic cancers) that have returned after a period of improvement (relapsed) after donor stem cell transplant. Immunotherapy with monoclonal antibodies, such as ipilimumab and nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum-tolerated dose (MTD) of ipilimumab or nivolumab administered to patients with relapsed hematologic malignancies following allogeneic stem cell transplantation. (Phase I) II. To characterize the toxicity of ipilimumab or nivolumab administered at the MTD in this patient population. (Phase Ib)

SECONDARY OBJECTIVES:

I. To assess response rate. II. To assess progression free and overall survival.

EXPLORATORY OBJECTIVE:

I. To assess the phenotypic and functional effects of ipilimumab or nivolumab on immune cells.

OUTLINE: This is a dose-escalation study.

INDUCTION PHASE: Patients receive ipilimumab intravenously (IV) over 90 minutes on day 1. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive nivolumab IV over 30 minutes on day 1. Treatment repeats every 14 days for 8 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE PHASE: Patients receive ipilimumab IV over 90 minutes. Treatment repeats every 12 weeks beginning at cycle 5 (24 weeks after the first dose of ipilimumab) for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients achieving clinical benefit will have the option to continue with ongoing maintenance dosing every 12 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive nivolumab IV over 30 minutes every 2 weeks in the absence of disease progression or unacceptable toxicity. Treatment repeats every 14 days for up to a total of 60 weeks (including Induction) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed hematologic malignancy
* The following malignancies will be considered eligible if progressive or persistent:

  * Chronic lymphocytic leukemia (CLL)
  * Non-Hodgkin lymphoma (NHL)
  * Hodgkin lymphoma (HL)
  * Multiple myeloma (MM)
  * Acute leukemia (acute myeloid leukemia [AML], acute lymphoblastic leukemia [ALL])
  * Myelodysplastic syndrome (MDS)
  * Myeloproliferative neoplasms (MPN)
  * Chronic myeloid leukemia (CML)
* Life expectancy of greater than 3 months
* Must have undergone allogeneic hematopoietic stem cell transplantation (HSCT) (regardless of stem cell source)
* Must have baseline donor T cell chimerism of >= 20%
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (unless due to Gilbert's disease or disease-related hemolysis, then =< 3.0 x ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x institutional ULN
* Creatinine =< 1.5 x institutional ULN
* Prednisone dose =< 5 mg/day and off all other systemic immunosuppressive medications for at least 4 weeks prior to study entry
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who have had anti-tumor therapy or other investigational agents within 4 weeks prior to registration (6 weeks for nitrosoureas or mitomycin C), or those who have not recovered from adverse events due to agents administered more than 4 weeks prior to registration
* Patients with prior history of or active severe (grade 3 or 4) acute graft-versus-host disease (GVHD)
* Patients with a history of prior treatment with ipilimumab, anti-programmed cell death protein 1 (PD 1) antibody, or cluster of differentiation (CD)137 agonist therapy are ineligible for the ipilimumab arm, but are eligible for the nivolumab arm
* Patients who have had donor lymphocyte infusion (DLI) within 8 weeks prior to registration
* Autoimmune disease: Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's disease, are excluded from this study, as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's granulomatosis]) and motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre syndrome and myasthenia gravis); patients with Hashimoto's thyroiditis are eligible to go on study
* Patients with known chronic human immunodeficiency virus (HIV), hepatitis B or hepatitis C infections should be excluded
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because ipilimumab and nivolumab are immunomodulatory agents with the potential for teratogenic or abortifacient effects; the effects of ipilimumab and nivolumab on the developing human fetus are unknown; for this reason and because immunomodulatory agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study or within 23 weeks after the last dose of study drug, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for at least 31 weeks after completion of ipilimumab or nivolumab administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2013-05-16 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of ipilimumab according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (Phase I) | At 12 weeks
  Dose-limiting toxic (DLT) effects were defined as grade III or IV acute graft versus host disease (GVHD), grade 4 hematologic toxic effects unrelated to the underlying disease, or grade 3 nonhematologic toxic effects that did not improve to grade 1 with a 3-week dose delay. Immune-related adverse events that resolved to grade 1 or lower with the use of glucocorticoids were not considered to be dose-limiting toxic effects. We designated the observation period for toxic effects to be 12 weeks to capture delayed immunologic toxic effects.
Maximum tolerated dose (MTD) of nivolumab according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (Phase I) | At 12 weeks
  Dose-limiting toxic (DLT) effects are defined as grade III or IV acute GVHD, grade 4 hematologic toxic effects unrelated to the underlying disease, or grade 3 nonhematologic toxic effects that did not improve to grade 1 with a 3-week dose delay. Immune-related adverse events that resolved to grade 1 or lower with the use of glucocorticoids were not considered to be dose-limiting toxic effects. We designated the observation period for toxic effects to be 12 weeks to capture delayed immunologic toxic effects.
Incidence of adverse events as assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (Phase Ib) | Up to 1 year after completion of study treatment
  A serious adverse event (SAE) is any adverse event, occurring at any dose and regardless of causality that 1) Results in death, 2) Is life-threatening, 3) Requires or prolongs inpatient hospitalization, 4) Results in persistent or significant disability/incapacity, 5) Is an important medical event when, based upon appropriate medical judgment, it may jeopardize the participant and require medical or surgical intervention to prevent one of the outcomes listed above.

SECONDARY OUTCOMES:
Clinical response | Up to 1 year
  Summarized by simple descriptive summary statistics delineating complete, partial, and best overall response, stable and progressive disease.
Progression-free survival (PFS) | From start of treatment to time of objective disease progression, assessed up to 1 year
  Using the Kaplan-Meier method. Will be analyzed and reported both for the entire cohort and within each disease group if feasible.
Overall survival (OS) | From the start of treatment to time of death, assessed up to 1 year
  Using the Kaplan-Meier method. Will be analyzed and reported both for the entire cohort and within each disease group if feasible.

OTHER OUTCOMES:
Change in immune cell numbers | Baseline to up to 1 year
  Laboratory studies will be performed to characterize the effects of ipilimumab and nivolumab in the post allogeneic stem cell transplantation (alloSCT) setting on B cells, NK, cells, or dendritic cells, both in terms of pre and post alloSCT changes in cell numbers.
Change in cytokine production | Baseline to up to 1 year
  Laboratory studies will be performed to characterize the effects of ipilimumab and nivolumab in the post alloSCT setting on B cells, NK, cells, or dendritic cells, both in terms of pre and post alloSCT changes in cell numbers.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew S Davids, Principal Investigator — Dana-Farber Cancer Institute
Locations (13):
- United States (13):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - City of Hope South Pasadena, South Pasadena, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Charlestown, Massachusetts

REFERENCES:
- [Derived] Penter L, Zhang Y, Savell A, Huang T, Cieri N, Thrash EM, Kim-Schulze S, Jhaveri A, Fu J, Ranasinghe S, Li S, Zhang W, Hathaway ES, Nazzaro M, Kim HT, Chen H, Thurin M, Rodig SJ, Severgnini M, Cibulskis C, Gabriel S, Livak KJ, Cutler C, Antin JH, Nikiforow S, Koreth J, Ho VT, Armand P, Ritz J, Streicher H, Neuberg D, Hodi FS, Gnjatic S, Soiffer RJ, Liu XS, Davids MS, Bachireddy P, Wu CJ. Molecular and cellular features of CTLA-4 blockade for relapsed myeloid malignancies after transplantation. Blood. 2021 Jun 10;137(23):3212-3217. doi: 10.1182/blood.2021010867. PMID 33720354
- [Derived] Davids MS, Kim HT, Costello C, Herrera AF, Locke FL, Maegawa RO, Savell A, Mazzeo M, Anderson A, Boardman AP, Weber A, Avigan D, Chen YB, Nikiforow S, Ho VT, Cutler C, Alyea EP, Bachireddy P, Wu CJ, Ritz J, Streicher H, Ball ED, Bashey A, Soiffer RJ, Armand P. A multicenter phase 1 study of nivolumab for relapsed hematologic malignancies after allogeneic transplantation. Blood. 2020 Jun 11;135(24):2182-2191. doi: 10.1182/blood.2019004710. PMID 32478814
- [Derived] Davids MS, Kim HT, Bachireddy P, Costello C, Liguori R, Savell A, Lukez AP, Avigan D, Chen YB, McSweeney P, LeBoeuf NR, Rooney MS, Bowden M, Zhou CW, Granter SR, Hornick JL, Rodig SJ, Hirakawa M, Severgnini M, Hodi FS, Wu CJ, Ho VT, Cutler C, Koreth J, Alyea EP, Antin JH, Armand P, Streicher H, Ball ED, Ritz J, Bashey A, Soiffer RJ; Leukemia and Lymphoma Society Blood Cancer Research Partnership. Ipilimumab for Patients with Relapse after Allogeneic Transplantation. N Engl J Med. 2016 Jul 14;375(2):143-53. doi: 10.1056/NEJMoa1601202. PMID 27410923